CLINICAL TRIAL: NCT00055393
Title: Bupropion Versus Placebo in the Treatment of Pathological Gambling
Brief Title: Bupropion in the Treatment of Pathological Gambling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Donald Black, Professor of and MD in Psychiatry, University of Iowa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 200007038; R21MH063289 (NIH); DSIR AT-AS
Record Dates: First submitted 2003-02-28; First posted 2003-03-03 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Pathological Gambling
MeSH Terms: conditions — Gambling | interventions — Bupropion

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

ARMS (2):
- Subjects receivng Bupropion (Active Comparator): The active arm subjects in this study (n = 18) received flexibly dosed bupropion in this randomized 12-week double-blind trial.
  Interventions: Drug: Bupropion
- Subjects receiving Placebo (Placebo Comparator): The inactive arm subjects in this randomly controlled study (n = 21) received a placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bupropion — 18 subjects in this randomly controlled double blind study received bupropion.
  Arms: Subjects receivng Bupropion
Drug: Placebo — 21 subjects received Placebo.
  Arms: Subjects receiving Placebo

SUMMARY:
This study will determine whether the drug bupropion is an effective treatment for Pathological Gambling.

DETAILED DESCRIPTION:
As gambling opportunities proliferate, PG has become a major health concern. Despite its importance, few treatment options with proven efficacy exist. This study will attempt to identify an effective treatment for PG.

Participants are randomly assigned to receive either bupropion or placebo for 12 weeks. Participants are assessed at baseline and at Weeks 2, 3, 4, 5, 6, 8, 10, and 12. Self administered questionnaires and interviews are used to assess participants. Follow-up assessments are made 1, 3, and 6 months after study completion.

ELIGIBILITY:
Inclusion Criteria:

* Meet the criteria for Pathological Gambling (DSM-IV-TR), through the administration of the National Opinion Research Center DSM Screen for Gambling Problems(NODS);
* Meet the criteria for Pathological Gambling (DSM-IV-TR), through the administration of the National Opinion Research Center DSM Screen for Gambling Problems(NODS);
* Receive a score of 5 or more on the South Oaks Gambling Screen (SOGS);
* Have PG for at least one year;
* Have had at least 2 or more gambling episodes during the 2-week screening period;
* Speak standard English;
* Be able to give written informed consent.

Exclusion Criteria:

* Evidence of current (past 3 months) substance misuse;
* Had a Hamilton Depression Rating Scale (HDRS)27 score of 18 or more (or a score on item 1 of greater than 2;
* Had a current eating disorder (except binge eating disorder);
* Had any history of seizures, or suicidal or aggressive behavior;
* Had a urine drug screen positive for stimulants, opiates, hallucinogens, or phencyclidine;
* Had a current or past psychotic disorder, bipolar disorder, or significant cognitive disorder;
* Received monoamine oxidase inhibitors within 3 weeks of randomization, long acting phenothiazine within 3 months of randomization,fluoxetine within 4 weeks of randomization, or other psychotropic drugs within 2 weeks of randomization;
* Had prior exposure to bupropion;
* Were engaged in individual, group, or couples psychotherapy during the 2 weeks before randomization, (except Gamblers Anonymous).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2002-07; Primary Completion 2005-05 (Actual); Study Completion 2006-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald W Black, MD, Principal Investigator — University of Iowa
Locations (1):
- Roy J. and Lucille A. Carver College of Medicine, University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data.

REFERENCES:
- [Result] Black DW, Arndt S, Coryell WH, Argo T, Forbush KT, Shaw MC, Perry P, Allen J. Bupropion in the treatment of pathological gambling: a randomized, double-blind, placebo-controlled, flexible-dose study. J Clin Psychopharmacol. 2007 Apr;27(2):143-50. doi: 10.1097/01.jcp.0000264985.25109.25. PMID 17414236